CLINICAL TRIAL: NCT02487355
Title: Pediatric Caudal Epidural Dexmedetomidine Enhances Postoperative Analgesia of Magnesium Sulphate and Quality of Caudal Anesthesia in Lower Abdominal Surgeries
Brief Title: Pediatric Caudal Dexmedetomidine Enhances Postoperative Analgesia of Magnesium Sulphate in Lower Abdominal Surgeries
Acronym: JASayed
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, jehan ahmed sayed, Associate Professor (Anesthesiology and Critical Care)- College of Medicine, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB000087123
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Pain, Postoperative
Keywords: dexmedetomidine; magnesium sulphate
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Magnesium Sulfate; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- group (MG) (Active Comparator): Magnesium sulfate 50 mg add to 1 ml/kg of 0.25%of bupivacaine
  Interventions: Drug: Magnesium Sulphate
- group (D) (Active Comparator): Dexmedetomidine 1 μg/ kg to add to 1ml/kg of 0.25%of bupivacaine
  Interventions: Drug: Dexmedetomidine
- group (MD) (Active Comparator): 50 mg magnesium sulfate and Dexmedetomidine 1 μg/ kg to add to 1ml/kg of 0.25%of bupivacaine
  Interventions: Drug: Dexmedetomidine + Magnesium Sulphate + Bupivacaine
- group (C) (Active Comparator): 1ml/kg of 0.25%of bupivacaine + 1 ml of normal saline
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 1 μg/ kg
  Arms: group (D)
Drug: Magnesium Sulphate — Magnesium Sulphate 50 mg
  Arms: group (MG)
Drug: Bupivacaine — 1ml/kg of 0.25%of bupivacaine
  Arms: group (C)
Drug: Dexmedetomidine + Magnesium Sulphate + Bupivacaine — Dexmedetomidine 1 μg/ kg + Magnesium Sulphate 50 mg + 1ml/kg of 0.25%of bupivacaine
  Arms: group (MD)

SUMMARY:
The study will conduct to compare the efficacy of Magnesium sulphate & dexmedetomidine used as adjuvants to bupivacaine in caudal block to provide intra-operative anesthesia as well as post -operative analgesia in pediatric patients.

DETAILED DESCRIPTION:
asdsd

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female children, ASA I and II,Aged 6 months to 6 years, , undergoing elective surgical procedures expected to last more than 90 min, and scheduled to receive general anesthesia combined with caudal extradural block

Exclusion Criteria:

* Allergy to local anesthetics,coagulation disorders, infection at site of injection, anatomic abnormalities and congenital anomalies like spina bifid, ASA III or higher, Parental refusal and the current use of Calcium Channel Blockers or Medication that may affect the neurologic system

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Time to first analgesic requirement | 24 hours
  The time from end of surgery to the first requirement of postoperative analgesia

SECONDARY OUTCOMES:
Postoperative sedation scores | 24 hours
  Level of sedation was recorded throughout the post-anesthesia care unit stay at 15-minute time intervals

CONTACTS AND LOCATIONS:
Overall Officials: jehan A Sayed, MD, Principal Investigator — assistant professor in anesthesia and intensive care department,faculty of medicine,Assiut univeristy,egypt
Locations (1):
- Assiut Univeristy Hospital, Asyut, Egypt